CLINICAL TRIAL: NCT02951286
Title: Skeletal and Dentoalveolar Changes Following Posterior Teeth Intrusion With High Pull Headgear in The Treatment of Patients With Anterior Open Bite
Brief Title: Molar Intrusion Using High Pull Headgear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-02-2016
Record Dates: First submitted 2016-10-28; First posted 2016-11-01 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Anterior Openbite
Keywords: Skeletal openbite; Molar intrusion; high pull headgear
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- high pull headgear + OBA (Experimental): A modified version of the Open Bite Appliance (OBA),introduced by Erverdi and Usumez, will be applied with high pull headgear for Orthoclassic ®1300 NE Alpha Drive, McMinnville, OR 97128 USA 866.752.0065.
  Interventions: Device: high pull headgear + OBA
- OBA (control group) (Experimental): A modified version of the Open Bite Appliance (OBA),introduced by Erverdi and Usumez, will be applied only.
  Interventions: Device: OBA (control group)

INTERVENTIONS:
Device: high pull headgear + OBA — a modified version of the OBA (Open Bite Appliance),introduced by Erverdi and Usumez, will be applied in compination with a high pull headgear.
  Arms: high pull headgear + OBA
Device: OBA (control group) — A modified version of the OBA (Open Bite Appliance),introduced by Erverdi and Usumez, will be applied alone (Control group)
  Arms: OBA (control group)

SUMMARY:
This prospective clinical study will evaluate the effect of high pull headgear for molar intrusion, compared with the control group, in adolescent patients with open bite malocclusion.

The study sample will consist of 24 patients with anterior open bite divided equally in two groups. The sample will be collected consecutively from patients attending the Orthodontic Department at Damascus university.

A modified version of the OBA (Open Bite Appliance),introduced by Erverdi and Usumez, will be applied for all patients. High pull headgears will be used in the first group, while, in the second (control) group, Open Bite Appliances will be used only.

The skeletal and dentoalveolar changes occurring after intrusion of posterior teeth will be assessed by using posteroanterior and lateral cephalometric radiographs; pre- and post- treatment changes for each group will be evaluated.

DETAILED DESCRIPTION:
Open bite malocclusion is considered one of the most difficult malocclusion to correct in orthodontic treatment because it appears as a result of different etiological factors such as genetic, dental, skeletal, functional, soft tissue, and habits that play roles in its development. Different treatment modalities used for the treatment of an anterior open bite. Multiloop edgewise archwires, miniscrews, high-pull headgear, and bite blocks have been used for anterior open bite patients, most open bite patients characterized by increased facial height, class II skeletal pattern, and vertical excess in maxillary posterior teeth.

Functional appliances, magnets, posterior bite blocks, and high pull headgear are used for posterior teeth intrusion. It is possible to generate intrusive force by using high pull headgear. Furthermore, direction of force can be changed according to the center of resistance of the dental units to achieve a better tooth movement control. The intrusion of posterior teeth will lead to decreased lower facial height by a counterclockwise rotation of the mandible; and improve class II skeletal relationship.

This study was the first clinical trial, that compare the effect of high pull headgear for molar intrusion with the control group in adolescent patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with skeletal open bite determined by an increased B angle (angle between maxillary plane and mandibular plane), sum of Bjork and the mandibular plane angle (angle between SN plane and mandibular plane).
* patients between 12 and 18 years old with permanent dentition stage.
* Negative over bite of more than a mm
* Class I and Class II skeletal anteroposterior relationship.

Exclusion Criteria:

* Previous orthodontic treatment.
* Patients with syndromes, clefts, or craniofacial abnormalities.
* Class III skeletal anteroposterior relationship.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Overbite | This variable will be evaluated twice; T0 before treatment, and T1 at the end of molar intrusion which will be abroximately after 7 months.
  The distance between the incisal edges of the upper and lower incisors, measured in mm.

SECONDARY OUTCOMES:
Molar intrusion | This variable will be evaluated twice; T0 before treatment, and T1 at the end of molar intrusion which will be approximately after 7 months
  The vertical distance between upper molars and the true horizontal plane (measured in mm)
Mandibular autorotation | This variable will be evaluated twice; T0 before treatment, and T1 at the end of molar intrusion which will be approximately after 7 months
  This variable will be measured by superimposition of the anterior cranial base
Anterior facial height | This variable will be evaluated twice; T0 before treatment, and T1 at the end of molar intrusion which will be approximately after 7 months
  The distance between the point "N" and the point "Me"
Change in the anteroposterior position of the point "B" | This variable will be evaluated twice; T0 before treatment, and T1 at the end of molar intrusion which will be approximately after 7 months
  The horizontal distance between point "B" and the true vertical plane

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Yousef, DDS MSc PhD, Study Director — Damascus University
Locations (1):
- Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No
The IPD will be available to all researchers in Damascus University

REFERENCES:
- [Result] Deguchi T, Kurosaka H, Oikawa H, Kuroda S, Takahashi I, Yamashiro T, Takano-Yamamoto T. Comparison of orthodontic treatment outcomes in adults with skeletal open bite between conventional edgewise treatment and implant-anchored orthodontics. Am J Orthod Dentofacial Orthop. 2011 Apr;139(4 Suppl):S60-8. doi: 10.1016/j.ajodo.2009.04.029. PMID 21435540
- [Result] Hart TR, Cousley RR, Fishman LS, Tallents RH. Dentoskeletal changes following mini-implant molar intrusion in anterior open bite patients. Angle Orthod. 2015 Nov;85(6):941-8. doi: 10.2319/090514-625.1. Epub 2014 Dec 22. PMID 25531420
- [Result] Lee J, Miyazawa K, Tabuchi M, Kawaguchi M, Shibata M, Goto S. Midpalatal miniscrews and high-pull headgear for anteroposterior and vertical anchorage control: cephalometric comparisons of treatment changes. Am J Orthod Dentofacial Orthop. 2013 Aug;144(2):238-50. doi: 10.1016/j.ajodo.2013.03.020. PMID 23910205